CLINICAL TRIAL: NCT06368687
Title: Anorexia Nervosa and Autism - a Care Location Adapted for Both Conditions
Brief Title: TRANPAS - TReating Anorexia Nervosa Plus Autism Spectrum
Acronym: TRANPAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-06112-01
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Anorexia Nervosa; Autism Spectrum Disorder
Keywords: anorexia nervosa; autism; pilot study; validation
MeSH Terms: conditions — Anorexia Nervosa; Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Pilot study. Ten consecutive patients with anorexia nervosa (AN) plus autism will be admitted to the autism care location at an inpatient ward for eating disorders. The planned period of care for each patient is 12 weeks. The patient will be assessed (including weight, height, self-report questionnaires and interviews) before admission, at discharge and 6 months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anorexia nervosa plus autism (Other): The treatment model takes into account the patient's perception disorders. This means e.g. an adapted mealtime situation where the patient can eat separately or wear hearing protection if necessary. The patients have an adapted meal plan regarding difficulties with specific textures or foods. To meet their need for continuity, they have the same contact persons throughout the entire period of care. The healthcare staff receive training in working with the specific subgroup and have regular exchanges of experience regarding the patient group, 15 minutes every or every two weeks.
  Interventions: Other: Anorexia nervosa plus autism

INTERVENTIONS:
Other: Anorexia nervosa plus autism — In the inpatient care the treatment model takes into account the patient's perception disorders, meaning e.g. an adapted mealtime situation where the patient can eat separately or wear hearing protection if necessary. The patients have an adapted meal plan regarding difficulties with specific textures or foods. To meet their need for continuity, they have the same contact persons throughout the entire period of care. The healthcare staff receive training in working with the specific subgroup and have regular exchanges of experience regarding the patient group, 15 minutes every or every two weeks.

SUMMARY:
In a pilot study, the investigators will validate a so-called autism care location in an inpatient ward. The care location will be adapted for patients with anorexia nervosa (AN) and concurrent autism (AN+autism). In order to investigate the effect of a tailored care location for patients with AN + autism, the evaluation will include weight development and changes in nutritional intake, eating disorder and anxiety symptoms. The overall aim is to improve treatment for this specific AN subgroup, that otherwise has a worse prognosis regarding AN recovery.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious eating disorder and has the highest mortality rate of all psychiatric illnesses. Adolescence is the most common age of onset. Nine out of ten people who fall ill are girls/women, and 2% of all girls/women will fall ill with AN at some point in their lives. In AN, one engages in self-starvation, which in turn leads to underweight. 75 - 80% of individuals with AN recover during adolescence, while the remainder are at high risk of developing chronic AN. For the individual, the chronic condition means great suffering in the form of serious psychiatric and somatic co-morbidity, social isolation and reduced/lack of work ability. People with autism show social withdrawal and reduced flexibility, reminiscent of the symptoms seen in AN. An estimated 15 - 20% of all individuals with AN also have autism. People with AN and concurrent autism run an increased risk of a worse prognosis, as they have more difficulty absorbing treatment, which in itself increases the risk of the condition becoming chronic. Today, there is no scientific evidence for how people with AN and concurrent autism should be treated.

In a pilot study, the investigators will validate a so-called autism care location in our inpatient ward, at Sahlgrenska University Hospital in Gothenburg, Sweden. The care location will be adapted for patients with AN and concurrent autism (AN+autism). In order to investigate the effect of a tailored care location for patients with AN + autism, the evaluation will include weight development and changes in nutritional intake, eating disorder and anxiety symptoms. The overall aim is to improve treatment for this specific AN subgroup, that otherwise has a worse prognosis regarding AN recovery.

ELIGIBILITY:
Inclusion Criteria:

* 25 years or older
* Meeting criteria for both anorexia nervosa and autism spectrum disorder according to the DSM-5
* In need of inpatient care due to anorexia nervosa

Exclusion Criteria:

* 24 years or younger
* Not in need of inpatient care due to anorexia nervosa
* Not meeting criteria for both anorexia nervosa and autism spectrum disorder according to the DSM-5

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
BMI change between baseline and discharge 12 weeks later | At admission, at discharge 12 weeks later, and 6 months after discharge
  Body Mass Index: weight (kilograms)/height (meters)2

SECONDARY OUTCOMES:
Change of level of anxiety between baseline and discharge 12 weeks later | At admission, at discharge 12 weeks later, and 6 months after discharge
  Anxiety assessed using General Anxiety Disorder 7-item (GAD-7)
Change of Quality of life between baseline and discharge 12 weeks later | At admission, at discharge 12 weeks later, and 6 months after discharge
  Quality of life (QoL) assessed using Short Form Health Survey (SF-36)